CLINICAL TRIAL: NCT01898130
Title: A Phase II Trial of Bevacizumab in Patients With Recurrent Solid Tumor Brain Metastases Who Have Failed Whole Brain Radiation Therapy
Brief Title: Bevacizumab in Pats w/ Recurrent ST Brain Metas Who Have Failed Whole Brain Radiation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 12C06; NCI-2013-00448 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00080404 (Other: Northwestern University IRB#)
Record Dates: First submitted 2013-06-28; First posted 2013-07-12 (Estimated); Results first posted 2019-04-25 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-03

CONDITIONS: Metastatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (bevacizumab) (Experimental): Patients receive bevacizumab IV over 30-90 minutes every 2 weeks. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Procedure: quality-of-life assessment

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This is a study to evaluate a drug called bevacizumab in patients with cancer whose disease has spread to their brain. This study will not evaluate the effect of bevacizumab on the systemic solid tumor cancer. Bevacizumab is a medication and it is thought that bevacizumab may interfere with the growth of new blood vessels; therefore it might stop tumor growth and possibly shrink the tumor by keeping it from receiving nutrients and oxygen supplied by the blood vessels.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the radiographic response rate in patients with solid tumor brain metastases treated with bevacizumab.

SECONDARY OBJECTIVES:

I. Estimate the progression-free survival (PFS) rate at 6 months. II. Determine the time to progression based on magnetic resonance imaging (MRI) or computed tomography (CT) scans.

III. Determine the time to response based on radiographic imaging. IV. Determine the duration of response based on radiographic imaging. V. Determine overall survival. VI. Collect additional safety data. VII. Assess changes in quality of life using the Functional Assessment of Cancer Therapy-Brain (FACT-Br) while on treatment.

OUTLINE:

Patients receive bevacizumab intravenously (IV) over 30-90 minutes every 2 weeks. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically or cytologically confirmed non-central nervous system (CNS) primary solid malignancy at the time of initial diagnosis; NOTE: brain lesions are not required to have pathologic confirmation; in addition, a copy of the pathology report for the primary tumor is sufficient for registration purposes
* Patients must have radiographically-confirmed recurrent brain metastases from a solid tumor after WBRT
* Patients must have measurable or evaluable disease in the brain
* Patients must have been on a stable dose of corticosteroids >= 5 days prior to obtaining their baseline gadolinium (Gd)-MRI of brain
* Patients must have completed WBRT > 12 weeks prior to enrollment to limit cases of pseudoprogression; however if new lesions are noted < 12 weeks but > 4 weeks prior to enrollment, those patients are eligible
* Patients who underwent radiosurgery to treat a progressive lesion must have confirmation of tumor by tissue, magnetic resonance spectroscopy (MRS), magnetic resonance (MR) perfusion or positron emission tomography (PET) and the lesion must be measurable; NOTE: radiosurgery may be done to a lesion that will not be used for response evaluation and should be done > 2 weeks prior to enrollment
* Patients may be on other systemic chemotherapies if progressive CNS disease occurs while on these treatments; NOTE: new systemic chemotherapies should not be started unless required to treat systemic disease and should not start until at least 1 follow up imaging study has been performed
* Patients may have received any number of prior CNS directed therapies - there are no limitations
* Patients must have a life expectancy of >= 12 weeks
* Patients must have a Karnofsky performance score (KPS) of >= 60
* Whole blood cell (WBC) >= 3,000/ul
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelets >= 100,000/mm^3
* Hemoglobin >= 10 gm/dl (may be reached by transfusion)
* Serum glutamic oxaloacetic transaminase (SGOT) < 2 x upper limit of normal (ULN) (or < 5 x ULN if liver is involved)
* Bilirubin < 2 x ULN (or < 5 x ULN if liver is involved)
* Creatinine < 1.5 x ULN
* Patients of both sexes must agree to the use of barrier contraceptives throughout the duration of treatment on this trial and for 3 months after discontinuing treatment; NOTE: hormonal contraceptives are not acceptable as a sole method of contraception
* Patients must be > 4 weeks from any major surgery
* Patients NOT on warfarin must have a prothrombin time (PT)/international normalized ratio (INR) < 1.4 within 14 days prior to registration

  * Patients on full-dose anticoagulants (e.g., warfarin or low molecular weight [LMW] heparin) must meet BOTH of the following criteria within 14 days prior to registration:

    * No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
    * In-range INR (between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of LMW heparin
* Female patients of child-bearing potential must have a negative pregnancy test within 14 days prior to registration
* Patients must be willing and able to comply with study and/or follow-up procedures
* Patients must sign an informed consent prior to registration and before undergoing any study-specific procedures indicating that they are aware of the investigational nature of this study

Exclusion Criteria:

* Patients with a diagnosis of intrathoracic lung carcinoma of squamous cell histology are not eligible for participation
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using barrier birth control methods, are not eligible for participation
* Patients must not have baseline proteinuria within 14 days prior to registration as demonstrated by either:

  * Urine protein: creatinine (UPC) ratio < 1.0 at screening, OR
  * Urine dipstick for proteinuria =< 2+; NOTE: patients discovered to have >= 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate =< 1g of protein in 24 hours to be eligible
* Patients must not have experienced any major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to registration, or be anticipated to need a major surgical procedure during the course of the study; NOTE: the exception is craniotomy
* Patients must not have experienced a core biopsy or other minor surgical procedure within 7 days prior to registration; NOTE: this excludes placement of a vascular access device
* Patients with a history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the previous 6 months are not eligible for participation
* Patients with a serious, non-healing wound, ulcer, or bone fracture are not eligible for participation due to the effects on vasculature by bevacizumab which may impair healing
* Patients known to be human immunodeficiency virus (HIV) or hepatitis B and/or C positive are not eligible for participation; NOTE: HIV and hepatitis testing is not required for study participation
* Patients with a history of any other cancer (except for non-melanoma skin cancer or carcinoma in-situ of the cervix), are not eligible for participation unless they are in complete remission and have been off of all therapy for that disease for a minimum of 3 years
* Patients receiving or participating on any other experimental agents/clinical trials are not eligible for participation
* Patients with a known hypersensitivity to any component of bevacizumab are not eligible for participation
* Patients with any significant medical illnesses or infection that, in the investigator's opinion, cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy are not eligible for participation
* Patients with leptomeningeal disease are not eligible for participation
* Patients who have received previous treatment with bevacizumab for CNS disease are not eligible for participation
* Patients with inadequately controlled hypertension (defined as systolic blood pressure > 150 and/or diastolic blood pressure > 100 mmHg) are not eligible for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-11-27 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2018-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priya Kumthekar, Principal Investigator — Northwestern University
Locations (4):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - Northwestern Memorial Hospital: Lake Forest Hospital, Lake Forest, Illinois
  - Cadence Health - CDH, Warrenville, Illinois
  - Columbia University Medical Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on October 11, 2013 with an accrual goal of up to 27 patients. The first patient started treatment November 27, 2013. The study was designed to enroll 9 patients initially and do an interim efficacy assessment. The study was closed permanently on April 24, 2017 with 27 patients enrolled.
Groups:
- Treatment (Bevacizumab): Patients receive 10mg/kg bevacizumab IV over 30-90 minutes every 2 weeks. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Bevacizumab: Given IV
  Quality-of-life assessment: Ancillary studies
Period: Treatment
Arm/Group | Treatment (Bevacizumab)
Started | 27
Reached 1st Response/2 Cycles | 24
Went on to Start Cycle 3 | 21
Completed | 21
Not Completed | 6
Not completed — Withdrawal by Subject | 2
Not completed — Progressive Disease | 4
Period: Follow up Until PD or Death
Arm/Group | Treatment (Bevacizumab)
Started | 27 (All patients treated on study go into follow up period for survival data.)
Completed | 26
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Bevacizumab)
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Objective Radiographic Tumor Response in Patients With Recurrent Solid Tumor Brain Metastases Treated With Bevacizumab
Description: Radiographic Response to treatment will be assessed prior to every odd-numbered cycle using CT or MRI scans until disease progression, unacceptable toxicity as assessed by the Response Assessment in Neuro-Oncology (RANO) Criteria for target lesions. Response is defined as the number of patients with Complete Response (CR) plus those with Partial Response (PR) radiographically. Generally CR is defined as the disappearance of all target lesions and PR is defined as >=50% decrease in the sum of the longest diameter of target lesions.
Time Frame: Every other cycle, starting cycle 3 (1 cycle =28 days) until off study. Range of cycles completed 1-20.
Population: Not all patients treated on study were determined to be evaluable for this objective as they did not receive follow up scans after the baseline scans.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Bevacizumab)
Number analyzed (Participants) | 24
Participants | 2

2. Secondary Outcome: Progression-Free Survival (PFS) at 6 Months in Patients With Recurrent Solid Tumor Brain Metastases Treated With Bevacizumab
Description: Progression-Free Survival (PFS) will be measured as the time from the first dose to the first occurrence of progression or death for any reason. To estimate PFS, Kaplan-Meier curves will be calculated and PFS at 6 months will be determined from the progression-free survival curve.
  Progression is defined using Response Assessment in Neuro-Oncology Criteria (RANO), as a 25% or more increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: At 6 months from treatment initiation.
Measure: Median (95% Confidence Interval); unit: percentage of patients with PFS
Arm/Group | Treatment (Bevacizumab)
Number analyzed (Participants) | 24
percentage of patients with PFS | 46 [25 to 67]

3. Secondary Outcome: Time to Progression in Patients With Recurrent Solid Tumor Brain Metastases Treated With Bevacizumab
Description: MRI or CT scans and clinical assessment will be used to measure Time to Progression which will be assessed as the time from the date of first dose to the date of first observation of progressive disease, non-reversible neurologic progression or increasing steroid requirements, or early discontinuation of treatment as assessed by the RANO Criteria in those patients that experience response.
Time Frame: From treatment initiation, every 2 cycles (1 cycle = 28 days) until progressive disease. Range of cycles completed 1-20.
Population: 6 patients experienced response and were evaluable for this outcome measure
Measure: Mean (Full Range); unit: Days
Arm/Group | Treatment (Bevacizumab)
Number analyzed (Participants) | 6
Days
  All Partial Response Patients | 300 [91 to 545]
  Clinical Partial Response: number analyzed (Participants) | 4
  Clinical Partial Response | 187 [91 to 314]
  Radiological Partial Response: number analyzed (Participants) | 2
  Radiological Partial Response | 525 [504 to 545]

4. Secondary Outcome: Time to Response in Patients With Recurrent Solid Tumor Brain Metastases Treated With Bevacizumab
Description: MRI or CT scans and clinical assessment will be used to measure Time to Response which will be assessed as the time from the date of first dose to the date of first observed tumor response in all patients that a response is observed. Response to treatment will be assessed using the Response Assessment in Neuro-Oncology (RANO) Criteria for target lesions. Response is defined as either Complete Response (CR) or a Partial Response (PR) radiographically. Generally CR is defined as the disappearance of all target lesions and PR is defined as >=50% decrease in the sum of the longest diameter of target lesions.
Time Frame: From the start of treatment every 2 cycles (1 cycle =28 days) until time of response. Range of cycles completed 1-20.
Population: 6 patients experienced a response and were therefore evaluable for this outcome measure.
Measure: Mean (Full Range); unit: Days
Arm/Group | Treatment (Bevacizumab)
Number analyzed (Participants) | 6
Days
  All Partial Response Patients | 73 [53 to 116]
  Clinical Partial Response: number analyzed (Participants) | 4
  Clinical Partial Response | 78 [53 to 116]
  Radiological Partial Response: number analyzed (Participants) | 2
  Radiological Partial Response | 62 [55 to 69]

5. Secondary Outcome: Duration of Response in Patients With Recurrent Solid Tumor Brain Metastases Treated With Bevacizumab
Description: The Duration of Overall Response is measured from the time measurement criteria are met for Complete Response (CR) or Partial Response (PR) until the first date that recurrent or Progressive Disease (PD) is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Duration of response will be based on CT or MRI scans and clinical assessment performed prior to every odd-numbered cycle to detect date of first response to study treatment until date of disease progression and assessed by the Response Assessment in Neuro-Oncology (RANO) Criteria for target lesions. Generally CR is defined as the disappearance of all target lesions, PR is defined as >=50% decrease in the sum of the longest diameter of target lesions and PD is defined as a 25% or more increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From documentation of response, every two cycles (1 cycle =28 days) until progressive disease. Range of cycles completed 1-20.
Population: Patients that achieved documented Complete Response or Partial Response were evaluated for this outcome measure
Measure: Mean (Full Range); unit: Days
Arm/Group | Treatment (Bevacizumab)
Number analyzed (Participants) | 6
Days
  All Partial Response Patients | 227 [11 to 490]
  Clinical Partial Response: number analyzed (Participants) | 4
  Clinical Partial Response | 110 [11 to 119]
  Radiological Partial Response: number analyzed (Participants) | 2
  Radiological Partial Response | 463 [435 to 490]

6. Secondary Outcome: Overall Survival (OS) in Patients With Recurrent Solid Tumor Brain Metastases Treated With Bevacizumab
Description: Overall Survival (OS) will be measured as the date of first dose of bevacizumab to the date of death from any cause. To estimate OS, Kaplan-Meier curves will be calculated and OS will be determined from the overall survival curve.
Time Frame: From start of treatment until death from any cause. Median follow up of 8 months (range 1.3 to 47.9 months)
Population: All patients included in OS outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Bevacizumab)
Number analyzed (Participants) | 27
Months | 8.2 [4.2 to 12.0]

7. Secondary Outcome: Toxicity of Bevacizumab in Patients With Recurrent Solid Tumor Brain Metastases
Description: Adverse events (AE) will be collected at the start of every cycle and graded according NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. All AEs that are determined to be grade 3 or higher and at least possible related to bevacizumab will be reported for toxicity. In general AEs will be graded:
  Grade 1 - Mild: the event causes discomfort without disruption of normal daily activities.
  Grade 2 - Moderate: the event causes discomfort that affects normal daily activities.
  Grade 3 - Severe: the event makes the patient unable to perform normal daily activities or significantly affects his/her clinical status.
  Grade 4 - Life-threatening: the patient was at risk of death at the time of the event.
  Grade 5 - Fatal: the event caused death.
Time Frame: Assessed prior to every cylcle (cycle=28 days) while on treatment through 30 days post last dose. Range of cycles 1-20.
Population: All patients that receive at least one dose of bevacizumab are considered to be evaluable for toxicity outcome measure.
Measure: Number; unit: participants
Arm/Group | Treatment (Bevacizumab)
Number analyzed (Participants) | 27
participants
  Lymphocyte Count Decreased | 1
  Headache | 1
  Hypertension | 3
  Thromboembolic Event | 1

8. Secondary Outcome: Quality of Life Assessments in Patients With Recurrent Solid Tumor Brain Metastases Treated With Bevacizumab
Description: Changes in quality of life will be evaluated using questionnaires (FACT-Br) at baseline (before treatment initiation) and at cycle 3.
  Four FACT scales were calculated. The higher the value the better the score, i.e., the better the quality of life perceived by patient.
  FACT-G (Fact General, possible range 0 - 108) BrCS (Brain Cancer Subscale, possible range 0 - 92) TOTAL (FACT-G + BrCS, possible range 0 - 200) TOI (Trial Outcome Index = Physical Well Being _ Functional Well Being +BrCS, possible range 0 - 148)
Time Frame: Baseline and at Cycle 3 (1 Cycle = 28 days).
Population: 12 patients completed quality of life questionnaires at baseline and Cycle 3 and therefore are evaluable for this outcome measure.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Treatment (Bevacizumab)
Number analyzed (Participants) | 12
score on a scale
  Baseline FACT-G | 83.0 [67.7 to 105.0]
  Baseline BrCS | 64.8 [46.0 to 87.0]
  Baseline TOTAL | 147.8 [124.3 to 189.0]
  Baseline TOI | 106.0 [77.0 to 139.0]
  Cycle 3 FACT-G | 75.9 [50.8 to 99.0]
  Cycle 3 BrCS | 62.8 [36.1 to 80.0]
  Cycle 3 TOTAL | 138.7 [93.8 to 178.0]
  Cycle 3 TOI | 99.4 [57.1 to 130.0]

9. Post Hoc Outcome: Response Rate in Patients With Recurrent Solid Tumor Brain Metastases Treated With Bevacizumab
Description: Response Rate is defined as all patients with Complete Response plus those with Partial Response as assessed by Response Assessment in Neuro-Oncology (RANO) Criteria of CT or MRI scans for target lesions combined with clinical assessment. Generally RANO Response definitions are as follows:
  CR is defined as the disappearance of all target lesions and PR is defined as >=50% decrease in the sum of the longest diameter of target lesions.
Time Frame: Every other cycle, starting cycle 3 (1 cycle =28 days) until off study. Range of cycles completed 1-20.
Population: 3 patients were determined not to be evaluable for response outcome measures as they did not get follow up scans after baseline scans.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Bevacizumab)
Number analyzed (Participants) | 24
Participants | 6

10. Post Hoc Outcome: Progression Free Survival (PFS) in Patients With Recurrent Solid Tumor Brain Metastases Treated With Bevacizumab
Description: Progression Free Survival (PFS) is measured from the time of treatment initiation until documentation of progressive disease or death from any cause. To estimate PFS, Kaplan-Meier curves will be calculated and PFS will be determined from the progression-free survival curve.
  Progression is defined using Response Assessment in Neuro-Oncology Criteria (RANO), as a 25% or more increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From treatment initiation and every two cycles (1 cycle = 28 days) until disease progression. Median follow up of 8 months (range 1.3 to 47.9 months).
Population: All patients evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Bevacizumab)
Number analyzed (Participants) | 27
Months | 4.3 [3.3 to 7.7]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the start of treatment, through 30 days post last treatment with patients being treated twice (every 14 days) in a 28 day cycle. Range of cycles completed 1-20.
Arm/Group | Treatment (Bevacizumab)
All-Cause Mortality (participants affected / at risk) | 24/27
Serious Adverse Events (participants affected / at risk) | 19/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Bevacizumab) (N=27)
Clinical Decline (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1 — Patient also experienced Nausea and Vomiting at time of event
Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Viral Gastroenteritis (Infections and infestations) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Transient Ischemic Attack (Nervous system disorders) | 1
Death due to Intracranial Hemorrhage (Nervous system disorders) | 1 — Patient also experienced depressed level of consciousness and headache during this event
Headache (Nervous system disorders) | 1 — Patient also with hypertension during this event
Pneumonia (Infections and infestations) | 1 — Patient also experienced urinary tract infection during this event
Viral Illness (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 1
Death NOS (Not otherwise specified) (General disorders) | 1
Seizure (Nervous system disorders) | 2
Dysarthria (Nervous system disorders) | 1
Colitis (Gastrointestinal disorders) | 1 — Patient acquired multifocal pneumonia during this hospitalization
Blood Bilirubin Increased (Investigations) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Radiation Enteritis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 — Patient also with hypoxia, pleural effusions and DVT during this event
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Bevacizumab) (N=27)
Anemia (Blood and lymphatic system disorders) | 14
Tinnitus (Ear and labyrinth disorders) | 2
Blurred Vision (Eye disorders) | 3
Constipation (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 5
Edema Limbs (General disorders) | 2
Fatigue (General disorders) | 13
Fever (General disorders) | 2
Gait Disturbance (General disorders) | 2
Pain (General disorders) | 4
Sinusitis (Infections and infestations) | 3
Urinary Tract Infection (Infections and infestations) | 3
Fall (Injury, poisoning and procedural complications) | 3
Activated Partial Thromboplastin Time Prolonged (Investigations) | 2
Alanine Aminotransferase Increased (Investigations) | 6
Alkaline Phosphatase Increased (Investigations) | 8
Aspartate Aminotransferase Increased (Investigations) | 13
Blood Bilirubin Increased (Investigations) | 6
Lymphocyte Count Decreased (Investigations) | 20
Neutrophil Count Decreased (Investigations) | 5
Platelet Count Decreased (Investigations) | 8
Weight Gain (Investigations) | 2
Weight Loss (Investigations) | 8
White Blood Cell Decreased (Investigations) | 11
Anorexia (Metabolism and nutrition disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 20
Hypoalbuminemia (Metabolism and nutrition disorders) | 21
Hypocalcemia (Metabolism and nutrition disorders) | 12
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 12
Hyponatremia (Metabolism and nutrition disorders) | 19
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2
Amnesia (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 4
Dysarthria (Nervous system disorders) | 2
Dysphasia (Nervous system disorders) | 3
Headaches (Nervous system disorders) | 6
Memory Impairment (Nervous system disorders) | 2
Peripheral Motor Neuropathy (Nervous system disorders) | 2
Paresthesia (Nervous system disorders) | 2
Delirium (Nervous system disorders) | 2
Hematuria (Renal and urinary disorders) | 2
Urinary Incontinence (Renal and urinary disorders) | 2
Urinary Frequency (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2
Palmar-Planar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT01898130/Prot_SAP_000.pdf